CLINICAL TRIAL: NCT04225728
Title: Rationale and Design of Ferric Polymaltose Hydroxide and Iron Sucrose Evaluation on Performance and Oxydative Stress in Patient With Iron deficIency and Stable Heart Failure Study
Brief Title: Evaluation on Performance and Oxydative Stress in Patient With Iron deficIency and Stable Heart Failure Study
Acronym: ERADAL-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CN NGANOU-GNINDJIO, MD, MSc (Other Government)
Responsible Party: Sponsor-Investigator, CN NGANOU-GNINDJIO, MD, MSc, Dr, Principal investigator, Yaounde Central Hospital
Organization: Yaounde Central Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERADAL-HF
Record Dates: First submitted 2019-04-02; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Chronic Heart Failure (CHF); Iron Deficiency
Keywords: oxidative stress; exercise tolerance; intravenous route (IV); intramuscular route (IM)
MeSH Terms: conditions — Iron Deficiencies | interventions — Ferric Oxide, Saccharated; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Iron sucrose IV arm (Active Comparator): Perfusion of diluted iron sucrose i.v. in two weeks. Half of the total dose at Day 0 and the other half at Day 14
  Interventions: Drug: Iron Sucrose IV
- Ferric polymaltose hydroxide complex IM arm (Active Comparator): Injection in two series, begin at Day 0 and the second at Day 14. In each series, we administered 300 mg of iron IM until reach half of the dose
  Interventions: Drug: Ferric polymaltose hydroxide complex IM
- Placebo arm (Placebo Comparator): 100 ml i.v. of normal saline administered at Day 0 and at day 14.
  Interventions: Other: Saline solution

INTERVENTIONS:
Drug: Iron Sucrose IV — Intervention will consisted of the administration for the IV route.
  -The IV route in two doses will be diluted bolus injection of iron or normal saline at day 0 and day 14.
  Other Names: Iron Sucrose injection
  Arms: Iron sucrose IV arm
Drug: Ferric polymaltose hydroxide complex IM — Intervention will consisted of the administration for the IM route. Drug will be given in two series of injection; the first series will began at day 0 and consist of administration of 300 mg of iron per day in intramuscular injection up to the half of the total dose and the second series will began at day 14 for the administration of the other half with the same scheme than the first.
  Other Names: Iron polymaltose hydroxide complex IM
  Arms: Ferric polymaltose hydroxide complex IM arm
Other: Saline solution — 100 ml i.v. of normal saline administered at Day 0 and at day 14.
  Other Names: Placebo intervention
  Arms: Placebo arm

SUMMARY:
ERADAL-HF is a double blinded, multi-centre, prospective, randomized, three arm study, enrolled ambulatory patients with chronic heart failure [New York Heart Association (NYHA) class II/III], with iron deficiency [defined as ferritin <100 ng/mL, or ferritin 100-300 ng/mL if transferrin saturation (TSAT) <20%] and haemoglobin (Hb) < 15 g/dL. Patients were randomized 1:1:1 to treatment into three arms: a first group treated with intravenous iron supplementation, a second treated by intramuscular iron supplementation and the third one which have received placebo. These patients were followed-up during a period of 04 weeks.

The aim of this study is to assess the short term effect of parenteral iron supplementation on exercise tolerance and oxidative stress in patients with stable chronic heart failure and iron deficiency

DETAILED DESCRIPTION:
ERADAL-HF is a double blinded, multi-centre, prospective, randomized, three arm study, enrolled ambulatory patients with chronic heart failure [New York Heart Association (NYHA) class II/III], with iron deficiency [defined as ferritin <100 ng/mL, or ferritin 100-300 ng/mL if transferrin saturation (TSAT) <20%] and haemoglobin (Hb) < 15 g/dL. Patients were randomized 1:1:1 to treatment into three arms: a first group treated with intravenous iron supplementation, a second treated by intramuscular iron supplementation and the third one which have received placebo. These patients were followed-up during a period of 04 weeks.

The aim of this study is to assess the short term effect of parenteral iron supplementation on exercise tolerance and oxidative stress in patients with stable chronic heart failure and iron deficiency in a sub-Saharan Africa. In addition, it will also try to evaluate its effectiveness using the intramuscular route and this with a simplified administration scheme.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with stable CHF (NYHA II/III functional class)
* Screening serum ferritin <100 ng/mL or 100-300 ng/mL with transferrin saturation <20%.
* Haemoglobin < 15 g/dl ;
* On optimal background therapy (as determined by the investigator) for at least 4 weeks with no dose changes of heart failure drugs during the last 2 weeks (with the exception of diuretics). In general, optimal pharmacological treatment should include an angiotensin-converting enzyme inhibitor or angiotensin II receptor blocker and a beta blocker unless contraindicated or not tolerated and diuretic if indicated.
* Subject must be capable of completing the 6MWT
* Before any study-specific procedure, the appropriate written informed consent must be obtained.

Exclusion Criteria:

* Subject has known sensitivity to any of the products to be administered during dosing.
* History of acquired iron overload.
* History of erythropoietin-stimulating agent, i.v. iron therapy, and/or blood transfusion in previous 6 weeks prior to randomization.
* Oral iron therapy at doses >100 mg/day in previous 1 week prior to randomization. Note: ongoing use of multivitamins containing iron <75 mg/day is permitted.
* Body weight ≤35 kg.
* Exercise training programme(s) in the 3 months prior to screening or planned in the next 6 months.
* Chronic liver disease (including active hepatitis) and/or screening alanine transaminase or aspartate transaminase above three times the upper limit of the normal range
* Subject will not be available for all protocol-specified assessments.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Variation in 6-minute walk test (6MWT) distance | 4 weeks
  Variation in 6MWT in meter distance from the baseline to week 4. By using pedometer

SECONDARY OUTCOMES:
Change in quality of life assessed by the Minnesota Living With Heart Failure Questionnaire (MLWHFQ) | 4 weeks
  Minnesota Living With Heart Failure Questionnaire score at Week 4 adjusted for baseline
Change in serum ferritin concentration | 4 weeks
  Change in serum ferritin concentration (micromol/l) level from baseline to week 4. By immunology
Change in serum concentration of anti-oxidant markers: Reduced Glutathione (micromol) | 4 weeks
  Change in serum concentration of anti-oxidant markers from baseline to week 4. By spectrophotometer
Change in serum concentration of oxidant marker: Malondialdehyde (micromol/l) | 4 weeks
  Change in concentration of oxidant marker from baseline to week 4. By spectrophotometer
Change in Left Ventricle Ejection Fraction by Simpson method | 4 weeks
  Change in Left Ventricle Ejection Fraction (%) by Simpson method on echocardiography from baseline to week 4
Cost-effectiveness by using the Incremental Cost-effectiveness Ratio (ICER) | 4 weeks
  Cost-effectiveness by using the ICER questionnaire between the IV and the IM route
Standard safety assessments | 4 weeks
  Standard safety assessments: adverse events by questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Chris Nadege NGANOU-GNINDJIO, MD, MAS, Principal Investigator — Yaounde Central Hospital
Locations (1):
- Yaounde Central Hospital, Cardiology department, Yaoundé, Cameroon